CLINICAL TRIAL: NCT05284617
Title: Exploratory Phase 2A, Double-blind, Placebo-Controlled, Dose Escalation Study to Determine the Safety, Tolerability, PD, and PK of HU6 for the Treatment of Subjects With Obese Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Exploratory Ph 2A, Double-Blind, Placebo-Controlled Dose Escalation Study of Safety, Tolerability, PD, & PK of HU6 for Subjects With Obese HFpEF
Acronym: HFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rivus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIV-HU6-2201
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Intervention Model Description: This is a Phase 2A, randomized, parallel-group, placebo-controlled, double-blind, within subject dose escalation trial with 3 dose levels of HU6 and placebo. Subjects will be randomized (1:1) either to HU6 or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment: HU6 Planned doses of HU6; N = 31 (Experimental)
  Interventions: Drug: HU6
- Placebo Comparator Non-active study drug N = 31 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HU6 — HU6 is being evaluated for its efficacy in improving cardiovascular function in obese subjects with HF with preserved ejection fraction (HFpEF).
  Arms: Active Treatment: HU6 Planned doses of HU6; N = 31
Drug: Placebo — Placebo
  Arms: Placebo Comparator Non-active study drug N = 31

SUMMARY:
This is a Phase 2A, randomized, parallel-group, placebo-controlled, double-blind, within subject dose escalation trial with 3 dose levels of HU6 and placebo. Subjects will be randomized (1:1) either to HU6 or placebo. Two dose levels will be administered in sequential order (150 mg daily followed by 300 mg daily), each for 20 days, to reach the third and highest dose of 450 mg daily if safety and tolerability are demonstrated at the lower 2 preceding doses. Administration of the 450 mg high dose will continue for a total of 94 days, with a safety follow-up visit within ~14 days of the last dose.

DETAILED DESCRIPTION:
This is a Phase 2A, randomized, parallel-group, placebo-controlled, double-blind, within subject dose escalation trial with 3 dose levels of HU6 and placebo. Subjects will be randomized (1:1) either to HU6 or placebo. Two dose levels will be administered in sequential order (150 mg daily followed by 300 mg daily), each for 20 days, to reach the third and highest dose of 450 mg daily if safety and tolerability are demonstrated at the lower 2 preceding doses. Administration of the 450 mg high dose will continue for a total of 94 days, with a safety follow-up visit within ~14 days of the last dose.

Subjects will be screened over a 40-day period to determine their eligibility based on specific history, physical, laboratory, and imaging evaluations as per the Schedule of Assessments. While a single screening clinical site visit is indicated, an additional visit may be necessary to complete the screening procedures due to scheduling issues. A number of these assessments will serve as the baseline prior to drug administration. A central laboratory will be used for all assessments, including MRI, DEXA, clinical blood/plasma measures, transthoracic echocardiography, and CPET.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, ≥40 years of age.
2. Competent to understand the information given in the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved Informed Consent Form (ICF) and must sign the form prior to the initiation of any study procedures.
3. Body mass index (BMI) ≥30 kg/m2;
4. Signs and symptoms of HF in the judgement of the Investigator, and meets the following disease severity criteria:

   a. KCCQ OSS ≤80; b. NYHA Classification Class II-III; c. Baseline peak VO2 ≤18 mL/kg/min for females or ≤20 mL/kg/min for males; d. Respiratory exchange ratio (respiratory quotient) (RER [RQ]) at baseline of >1.0; e. Left ventricular ejection fraction (EF) ≥50%; f. At least 1 of the following objective criteria for HF: i. Documented hospitalization with HF as primary cause within in last year, or if greater than the past year, then with addition of structural heart disease on echocardiography (increased left atrial volume size or left ventricular hypertrophy, with sex-specific cut-points as per Lang, 2015) as follows:
   * Left ventricular hypertrophy (LVH):

     1. Men: Either septal wall thickness (cm) either ≥1.1 or posterior wall thickness ≥1.1;
     2. Women: Either septal wall thickness (cm) either ≥ 1.0 or posterior wall thickness ≥1.0;
   * Left atrial dilation (LAD): AP dimension (cm): ≥4.0 in men; >3.8 in women; ii. Pulmonary capillary wedge pressure (PCWP) at rest >15 mmHg (or left ventricular end-diastolic pressure [LVEDP] ≥18 mmHg) or >25 mmHg (or 2.0 mmHg/L/min) with exercise in the last year; iii. E/e' ratio ≥14 at septal annulus at rest on Doppler and tissue Doppler imaging in the last year; or iv. Currently elevated NT-proBNP defined as >125 pg/mL without atrial fibrillation and >350 pg/mL for subjects with chronic controlled atrial fibrillation.
5. Participants should maintain their stable level of physical activity throughout the duration of the study and must agree to not enroll in an exercise training program during the study.
6. Participants should maintain their stable diet and no plan to enter into a weight loss program prior to or during the course of the study.
7. Euthyroid as assessed by a thyroid profile utilizing thyroid stimulating hormone (TSH) and free thyroxine (T4) testing at screening. Subjects with a stable history of thyroid disease and who have been on stable doses of thyroid medications for a minimum of 4 months can be enrolled.
8. Ambulatory (not wheelchair- or scooter-dependent) and able to perform upright exercise testing including a 6 MWT.
9. Stable doses of medications (defined as no new medication or change in existing dose of medication ≥50%) for 30 days prior to screening, with additional specific criteria for the diuretics:

   1. If treated with a loop or thiazide diuretic, must be on stable regimen, which dose permits a flexible diuretic dosing schedule.

Exclusion Criteria:

1. Life expectancy <1 year due to non-cardiovascular reasons, in the judgement of the Investigator.
2. History of malignancy within 5 years (except non-high-grade skin cancers, carcinoma-in-situ, or low-grade prostate cancer).
3. Weight change (gain or loss) of ≥10 pounds either by self-reporting or documented weight loss within the past 90 days.
4. Bariatric surgery prior to screening or planned bariatric surgery during the course of the study.
5. Treatment with GLP-1 receptor antagonist begun within 1 year of screening.
6. Treatment with SGLT2 inhibitors begun within 6 months of screening.
7. Intolerance to MRI or with conditions contraindicated for MRI procedures including but not limited to:

   1. Having surgical clips/metallic implants/shrapnel/internal electric implants; or
   2. Inability to fit into MRI scanner due to subject habitus or exceeding weight tolerance limit of the scanner (generally, 350 or 400 lbs, dependent on manufacturer); or
   3. Claustrophobia: history of severe claustrophobia that would lead to inability to conduct MRI.
8. Current acute decompensated HF requiring intravenous (IV) diuretics or recent (<1 month before screening) hospitalization for HF.
9. Primary cardiomyopathy (e.g., constrictive, restrictive, infiltrative, toxic, hypertrophic [congenital], congenital, or any other primary cardiomyopathy, in the judgement of the Investigator.
10. Active myocarditis (COVID-induced or otherwise).
11. Active collagen vascular disease.
12. Current greater than moderate left- or right sided valve disease, in the opinion of the Investigator.
13. Planned cardiac surgery or catheter intervention during the time of trial participation.
14. Prior documented EF <40% within the last 3 years.
15. Tachycardia (>110 beats/minute) at screening.
16. Atrial fibrillation or atrial flutter with an uncontrolled heart rate response or with a resting heart rate greater than 110 bpm by ECG at screening. Subjects may rescreen after appropriate adjustment of medication to manage the atrial fibrillation. A maximum of 16 subjects with this condition can be enrolled in this study.
17. Untreated, life-threatening dysrhythmia.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluate weight reduction while on HU6 treatment | 5 months
  Assess the rate and amount of body weight loss over the course of HU6 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shaharyar Khan, PhD, Study Director — Rivus Pharmaceuticals, Inc.
Locations (15):
- United States (15):
  - National Heart Institute, Beverly Hills, California
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California
  - New Generation of Medical Research, Hialeah, Florida
  - Broward Research Center, Pembroke Pines, Florida
  - Northwestern University, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Mid America Heart Institute, Kansas City, Missouri
  - Weill Cornell Medicine, New York, New York
  - Wake Forest, Winston-Salem, North Carolina
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern, Dallas, Texas

REFERENCES:
- [Derived] Pandey A, Lewis GD, Borlaug BA, Shah SJ, Sauer AJ, Litwin S, Sharma K, Jorkasky DK, Tarka EA, Khan SM, Kitzman DW. Novel Controlled Metabolic Accelerator for Obesity-Related HFpEF: The HuMAIN-HFpEF Randomized Clinical Trial. JAMA Cardiol. 2025 Jun 1;10(6):609-616. doi: 10.1001/jamacardio.2025.0103. PMID 40072462